CLINICAL TRIAL: NCT02266966
Title: Effect of F2695 on Brain Activity Measured by Functional Magnetic Resonance Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F02695LP105
Record Dates: First submitted 2014-09-19; First posted 2014-10-17 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2013-12

CONDITIONS: Subject

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- F2695 (Experimental): Single dose - 2 capsules / Day on Day 1 and Day 8
  Interventions: Drug: F2695
- placebo (Placebo Comparator): Single dose - 2 capsules / Day on Day 1 and Day 8
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: F2695
  Arms: F2695
Drug: Placebo
  Arms: placebo

SUMMARY:
The aim of this functional Magnetic Resonance Imaging (MRI) study is to assess the effect of single dose of F2695 at 75mg on modulation of the cerebral motor network.

ELIGIBILITY:
Inclusion Criteria:

Male right-handed*, healthy volunteers 18 to 40 years of age. Having signed and dated an informed consent form

Exclusion Criteria:

Any significant disease or history of any clinically important drug allergy. Acute disease state within 7 days. History of drug abuse within 1 year. History or current excessive use of alcohol and / or positive alcohol screen. History of narrow angle glaucoma, seizures or epilepsy or brain injury. History of Gluten sensitivity, Gluten intolerance (celiac disease), Wheat allergy or Wheat intolerance.

History of obstructive voiding symptoms, including urinary retention.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Motor system cortical areas activation magnitude during a paced motor task. | 1 day (Period 1/Day +1, Period 2/Day +8)
  1. Location coordinates (x,y,z),
  2. Voxel cluster size expressed in terms number of voxels,
  3. Intensity as measured with a Z-score

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) as a measure of safety and tolerability | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: François Chollet, Principal Investigator — Hôpital Purpan CHU TOULOUSE, France
Locations (1):
- Centre d'Investigation Clinique (CIC), Toulouse, France